CLINICAL TRIAL: NCT04465201
Title: Advanced Impella® SmartAssist® System for Patient Monitoring & Treatment: The Smart Pump Study
Brief Title: The Smart Pump Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VV-TMF-16540
Record Dates: First submitted 2020-06-15; First posted 2020-07-10 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects receiving the Impella/Impella® Hemodynamics platform (Experimental)
  Interventions: Device: Impella CP with Smart Assist (Circulatory Support System)

INTERVENTIONS:
Device: Impella CP with Smart Assist (Circulatory Support System) — Subjects will receive the Impella® with the Impella® Hemodynamics Platform prior to High risk percutaneous coronary intervention (HRPCI). Device escalation or early termination of the study will be allowed for subjects as deemed necessary by the treating physician. Subjects will be consented for follow-up through discharge from the index HRPCI admission.

SUMMARY:
To demonstrate that the Impella® Hemodynamic Platform (the "Study Device") is safe, and measurements obtained are as good as currently used methods. These measurements include how much pressure the heart is generating and how much blood your heart is pumping during the PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Subject presents for elective PCI
3. Subject or the subject's LAR has signed the informed consent
4. Subject indicated for Impella® support

Exclusion Criteria:

1. Any contraindication or inability to place an Impella® including tortuous vascular anatomy, femoral bruits or absent pedal pulses
2. Cardiogenic shock defined as systemic hypotension (SBP<90mmHg or the need for inotropes/vasopressors to maintain an SBP >90mmHg) plus one of the following:

   1. Any requirement for inotropes/vasopressors prior to arrival at the catherization lab
   2. Clinical evidence of end organ hypoperfusion
   3. Use of IABP or any other circulatory support device
3. Suspected systemic active infection
4. Suspected or known pregnancy
5. Known contraindication to heparin, pork, pork products, or contrast media
6. Subject has other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures
7. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary end point.
8. Subject belongs to a vulnerable population [Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The ability to calculate and display cardiac output (CO). | Through study completion, approximately 2 days
  Defined as the number of times a CO calibration sequence is successfully completed and the CO is displayed divided by the number of times the pinging sequence is attempted. The endpoint is a rate and therefore has no units of measure. It is the "number of times CO was successfully completed, and CO is displayed" divided by the "number of times the pinging sequence was attempted"

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No